CLINICAL TRIAL: NCT07250412
Title: The Accuracy Of 3D Color Ultrasonography for Detecting the Degree of Placenta Accreta Spectrum Invasion
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Atef Ahmed, The Accuracy Of 3D Color Ultrasonography for Detecting the degree of placenta Accreta spectrum invasion, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-med-25-8____12MS
Record Dates: First submitted 2025-09-30; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-09

CONDITIONS: Placenta Accrete Spectrum
MeSH Terms: interventions — Cesarean Section

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasonography (Active Comparator)
  Interventions: Procedure: Cesarian section

INTERVENTIONS:
Procedure: Cesarian section — Cesarian section for detection the degree of placenta Accreta spectrum invasion comparaple to 3D color Doppler

SUMMARY:
To evaluate the correlation between preoperative ultrasound imaging findings by 3D Color Doppler Ultrasound and the intraoperative severity of Placenta Accreta Spectrum (PAS) disorders, in order to assess the diagnostic accuracy of sonographic markers and their utility in predicting the extent of placental invasion.

ELIGIBILITY:
Inclusion Criteria: Pregnant women with clinical or ultrasound suspicion of PAS, including:

1. Placenta previa or low-lying placenta
2. History of previous cesarean section(s) or uterine surgery (e.g., myomectomy, D&C) 2. Gestational age ≥ 28 weeks at the time of ultrasound evaluation 3. Undergoing planned cesarean delivery in the study hospital 4. Availability of preoperative ultrasound imaging performed using a standardized protocol.

   5. Patient can provide informed Written consent and Agree to participate in the study

   -

   Exclusion Criteria: Patients with incomplete or poor-quality ultrasound data 2. Unavailability of intraoperative confirmation of placental invasion 3. Patients with placental abruption or other causes of acute bleeding requiring emergency delivery without imaging 4. Loss to follow-up prior to delivery 5. Declined consent or withdrew participation from the study

   -

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between preoperative ultrasound findings and the confirmed degree of Placenta Accreta Spectrum (PAS) severity (classified as accreta, increta, or percreta). o The classification will be based on intraoperative surgical findings. | Patient preg 28 wks compare finding intraoperative
Correlation between preoperative ultrasound findings and the confirmed degree of Placenta Accreta Spectrum (PAS) severity (classified as accreta, increta, or percreta). o The classification will be based on intraoperative surgical findings. | Pt preg for more than 28wks preg and compare finding intraoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medecine Sohag university, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided